CLINICAL TRIAL: NCT06738953
Title: Preventing Mental Disorders in Young Adults with Low Self-efficacy: a Randomized Controlled Trial
Brief Title: Prevention of Mental Disorders Through Self-efficacy Interventions
Acronym: SELFTIE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Health and Medical University Potsdam (Other)
Collaborators: German Research Foundation (Other); Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Prof. Dr. Eva Asselmann, Prinicipal Investigator, Professor of Differential and Personality Psychology, Health and Medical University Potsdam
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: GEPRIS:534641939
Record Dates: First submitted 2024-11-21; First posted 2024-12-18 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Depression Disorders; Affective Disorders; Prevention; Substance Use Disorders; Self-Efficacy
Keywords: Prevention; Transdiagnostic; Young Adults; Online Intervention; Mental Health; Self-Efficacy; Depressive Disorders; Anxiety Disorders; Substance Use Disorders
MeSH Terms: conditions — Mood Disorders; Substance-Related Disorders; Psychological Well-Being; Depressive Disorder; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Selective Preventive Intervention Study
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Behavioral: Cognitive-behavioral intervention to increase self-efficacy (Experimental): n = 189 participants will be allocated randomly to this study arm.
  Interventions: Behavioral: Cognitive-Behavioral Intervention to increase Self Efficacy
- Behavioral: Group Discussion on Psychological Experiments as active Control (Placebo Comparator): n = 189 participants will be allocated randomly to this study arm.
  Interventions: Behavioral: Placebo: Weekly Recap and Group Discussion on Psychological Experiments

INTERVENTIONS:
Behavioral: Cognitive-Behavioral Intervention to increase Self Efficacy — Participants in the intervention group will receive a brief (6 sessions of 75-90 min each) cognitive-behavioral intervention. The intervention will be delivered in an online group format (subgroups of 8-12 participants). The courses will be structured according to well-established self-efficacy interventions with proven effectiveness (Bresó et al., 2011; Cieslak et al., 2016; Luszczynska et al., 2007), targeting Bandura's four key sources of self-efficacy (i.e., mastery experience, vicarious experience, verbal persuasion, and physiological/emotional arousal). Each session will consist of a theoretical and a practical part and be structured as follows: opening, discussion of homework (with special emphasis on participants' progress and sharing of experiences), introduction to the topic, practice, answering open questions, closing. The course sessions are accompanied by weekly homework assignments to be completed at home.
  Arms: Behavioral: Cognitive-behavioral intervention to increase self-efficacy
Behavioral: Placebo: Weekly Recap and Group Discussion on Psychological Experiments — Participants in the control group will meet in small groups (8-12 participants per group; 6 sessions, similar to the intervention group). They will receive a brief introduction to well-known psychological experiments and findings (e.g., the Asch experiment, selective attention) and discuss their perspectives on these topics, including personal implications of the experiments. Content related to self-efficacy or cognitive-behavioral interventions will be explicitly avoided. To prevent expectancy effects and other biases, participants will not be informed that they are part of the control group. If suspicions arise, participants will be told that group leaders are not allowed to disclose this. Group sessions will be led by a psychologist. The course materials (workbook, slides, and course instructions) will be shared on OSF.
  Arms: Behavioral: Group Discussion on Psychological Experiments as active Control

SUMMARY:
Low self-efficacy is a transdiagnostic risk factor for several mental disorders. Self-efficacy refers to one's belief that one is capable of performing a behavior necessary to successfully complete a task or achieve a goal. Consistent with theoretical models and empirical findings, individuals with low self-efficacy are more likely to perceive challenges as uncontrollable and threatening and thus are at increased risk for developing mental disorders during sensitive periods such as young adulthood. Self-efficacy interventions have been shown to be effective in promoting health behavior change, quality of life, and treatment adherence in patients with serious illnesses, as well as motivation and performance in students and employees. However, whether targeted self-efficacy training can prospectively prevent the onset of full-threshold anxiety, affective, and substance use disorders in young adults at increased risk for psychopathology remains an open question.

The aim of this randomized controlled trial is to test whether a brief cognitive-behavioral intervention in young adults with low self-efficacy can increase general self-efficacy (primary outcome of intervention effectiveness) and thus prevent the onset of DSM-5 mental disorders in the subsequent year (primary outcome of prevention effectiveness). In addition, we examine whether improvements in domain-specific self-efficacy lead to subsequent improvements in general self-efficacy and thus to lower psychopathological symptoms (spillover effects).

Young adults (18-30 years) with low self-efficacy but no mental disorder will be included (N=378). The study will include screening, entry, baseline, post, and 12-month follow-up assessments plus additional course assessments in both groups. After the baseline assessment, participants will be randomized to an intervention or control group. The intervention group will receive group-based self-efficacy training (6 sessions of 75-90 minutes each). The control group will also meet in groups (6 sessions) but will only talk about psychological research findings unrelated to self-efficacy or cognitive-behavioral interventions without receiving any training. DSM-5 mental disorders will be assessed at study entry and follow-up with a structured diagnostic interview. Other outcomes will be assessed with established scales and ecological momentary assessments (EMA) at baseline, post and follow-up. Clinical outcomes include psychopathological symptoms (dimensional scores for anxiety, depression, anger, and somatic symptoms, as well as sleep disturbance) and mental disorders (DSM-5 categorical diagnoses of anxiety, affective, and substance use disorders). Intervention effectiveness will be tested using logistic/linear regression and multilevel analyses. Spillover effects between improvements in domain-specific/general self-efficacy and psychopathological symptoms over the course of the study will be examined using cross-lagged panel models.

DETAILED DESCRIPTION:
Low self-efficacy is a transdiagnostic risk factor for several mental disorders. Self-efficacy refers to one's belief that one is capable of performing a behavior necessary to successfully complete a task or achieve a goal. Consistent with theoretical models and empirical findings, individuals with low self-efficacy are more likely to perceive challenges as uncontrollable and threatening and thus are at increased risk for developing mental disorders during sensitive periods such as young adulthood. Self-efficacy interventions have been shown to be effective in promoting health behavior change, quality of life, and treatment adherence in patients with serious illnesses, as well as motivation and performance in students and employees. However, whether targeted self-efficacy training can prospectively prevent the onset of full-threshold anxiety, affective, and substance use disorders in young adults at increased risk for psychopathology remains an open question.

The aim of this randomized controlled trial is to test whether a brief cognitive-behavioral intervention in young adults with low self-efficacy can increase general self-efficacy (primary outcome of intervention effectiveness) and thus prevent the onset of DSM-5 mental disorders in the subsequent year (primary outcome of prevention effectiveness). In addition, the investigators examine whether improvements in domain-specific self-efficacy lead to subsequent improvements in general self-efficacy and thus to lower psychopathological symptoms (spillover effects).

Young adults (18-30 years) with low self-efficacy but no mental disorder will be included (N=378). The study will include screening, entry, baseline, post, and 12-month follow-up assessments plus additional course assessments in both groups. After the baseline assessment, participants will be randomized to an intervention or control group. The intervention group will receive group-based self-efficacy training (6 sessions of 75-90 minutes each). The control group will also meet in groups (6 sessions) but will only talk about psychological research findings unrelated to self-efficacy or cognitive-behavioral interventions without receiving any training. DSM-5 mental disorders will be assessed at study entry and follow-up with a structured diagnostic interview. Other outcomes will be assessed with established scales and ecological momentary assessments (EMA) at baseline, post and follow-up. Clinical outcomes include psychopathological symptoms (dimensional scores for anxiety, depression, anger, and somatic symptoms, as well as sleep disturbance) and mental disorders (DSM-5 categorical diagnoses of anxiety, affective, and substance use disorders). Intervention effectiveness will be tested using logistic/linear regression and multilevel analyses. Spillover effects between improvements in domain-specific/general self-efficacy and psychopathological symptoms over the course of the study will be examined using cross-lagged panel models.

Detailed Description Based on previous research, it is plausible that self-efficacy training may have positive mental health effects and thus successfully prevent the development of mental disorders over time: Consistent with social cognitive theory, self-efficacy training may reduce feelings of anxiety and thus reduce the risk of anxiety disorders. According to the theory of learned helplessness, self-efficacy training may reduce feelings of helplessness and depression and thus reduce the risk of affective disorders. In addition, and consistent with the self-medication hypothesis, individuals who receive self-efficacy training may be less likely to use tobacco, alcohol, or medication/illicit drugs to avoid or down-regulate unpleasant feelings, thereby reducing the risk of substance use disorders.

However, although self-efficacy interventions have been shown to be beneficial in other domains, it remains unclear whether self-efficacy training can effectively prevent the onset of full-threshold anxiety, affective, and substance use disorders in young adults. Given that selective and indicated prevention has been shown to be particularly effective in high-risk samples young adults with low self-efficacy and thus increased risk for mental disorders may benefit from targeted self-efficacy training.

Study aims

This randomized controlled trial in young adults (aged 18-30 years) with low self-efficacy but no 12-month mental disorder at study entry aims to test whether a short cognitive-behavioral intervention in young adults with low levels of self-efficacy (but no 12-month anxiety, affective, or substance use disorder, current intervention (seeking) or suicidality) can effectively increase self-efficacy and thus prospectively prevent the onset of DSM-5 anxiety, affective, and substance use disorders in the subsequent year. The following hypotheses will be tested (based on screening, entry, baseline, post, and 12-month follow-up assessments plus additional course assessments in both groups:

Hypotheses

1. Participants in the intervention vs. control group experience a greater increase in general self-efficacy from baseline to post (primary outcome of intervention effectiveness) and greater improvements in dimensional psychopathological symptoms and other dimensional outcome measures from baseline to post (secondary outcome of intervention effectiveness). Note: Other dimensional outcome measures include self-esteem, perceived control, social support, coping strategies, interpersonal competence, work engagement, and individual work performance.
2. Participants in the intervention vs. control group experience a lower risk of incident DSM-5 mental disorders from entry to follow-up (primary outcome of prevention effectiveness) and greater improvements in dimensional psychopathological symptoms and other dimensional outcome measures from baseline to follow-up (secondary outcomes of prevention effectiveness). Note: Not only binary diagnoses but also dimensional symptoms will be assessed to be able to examine more nuanced symptom changes as well as lagged effects between changes in self-efficacy and changes in mental health over time.
3. In the intervention group, improvements in domain-specific self-efficacy will lead to subsequent improvements in general self-efficacy over the course of the intervention (i.e., week 1-6 of the training; spillover hypothesis 1). Note: In the intervention group, participants choose to work on their self-efficacy in the domains of health, social relationships, or education/work. In these analyses, domain-specific self-efficacy refers to the domain that the particular participant works on during the intervention. The selected domains are recorded systemically.
4. In the intervention group, improvements in general self-efficacy will lead to subsequent improvements in dimensional symptom outcomes over the course of the study (i.e., from baseline to follow-up; spillover hypothesis 2).

Design The investigators will conduct a randomized controlled trial (in young adults aged 18-30 years with low levels of general self-efficacy but no 12-month anxiety, affective, or substance use disorder, current intervention (seeking), or suicidality with an intervention group and a control group. Participants in the intervention group will receive group-based self-efficacy training (8-12 participants per group; 6 sessions of 75-90 minutes each). Participants in the control group will also meet in groups (8-12 participants per group; 6 sessions) but will only talk about psychological research findings unrelated to self-efficacy or cognitive-behavioral interventions without receiving any training. The design contains three measurement points at which the main outcome variables self-efficacy and psychopathology are assessed: 1) a baseline assessment - immediately before the courses; 2) a post-assessment - immediately after the courses; 3) a 12-month follow-up assessment - 12 months after the post-assessment.

Procedure Individuals who meet the inclusion criteria will participate in the baseline assessment. After the baseline assessment, participants will be randomized to either the intervention or control group. Before each course session (6 times), both general and domain-specific self-efficacy will be assessed. Dimensional clinical outcomes will be measured at baseline, post-intervention, and at a 12-month follow-up. Additionally, a one-week EMA will be administered at these three time points.

The intervention will be delivered in an online group format (subgroups of 8-12 participants; 6 sessions of 75-90 minutes each) and led by a psychologist. The courses will be structured according to well-established self-efficacy interventions with proven effectiveness, targeting Bandura's 4 key sources of self-efficacy (i.e., mastery experience, vicarious experience, verbal persuasion, and physiological/emotional arousal).

Course sessions will be structured as follows: Opening, brief reflection on current progress toward the goal, discussion of homework (with special emphasis on participants' progress and sharing of experiences), introduction to the topic, supervised practice, answering open questions, and closing. Course sessions will be accompanied by weekly homework assignments for practice at home. Assignments will be prepared and discussed during each class session. Participants will also be asked to keep a homework and success diary (workbook) to document changes in thoughts, feelings and behaviors, questions/difficulties (to be discussed in the next session), and accumulating successes in daily life over time (to enhance vicarious experiences).

To increase adherence to the intervention, participants will receive a weekly text message with homework reminders and motivational support. Participants in the intervention group will be able to contact a psychologist between sessions to ask questions and receive additional support regarding the intervention and homework. The intervention will be tested in a pilot phase in which self-efficacy will be measured before, during, and after the intervention. In addition, feedback interviews on the intervention will be conducted during the pilot phase to assess its acceptability, and the intervention will be modified accordingly if needed.

Recruitment Participants will be recruited through personal contact and print/online advertisements in universities and vocational schools, businesses, coworking spaces, clubs, bars, cafes, restaurants, cinemas, theaters, fitness centers and sports clubs, pharmacies, general practitioners, health insurance companies, and public and social media. Recruitment sites will also include social and welfare institutions that cater to individuals from diverse backgrounds (e.g., low education or migration) to ensure an inclusive sample and to counteract common biases in intervention research (e.g., overrepresentation of highly educated groups). Participants will be recruited not only in Berlin and Potsdam, but also in other (metropolitan and rural) regions of Germany and via online media.

Inclusion and exclusion criteria are listed below. After the baseline examination, individuals who meet the inclusion criteria will participate in the baseline examination. After the baseline assessment, they will be randomized to the intervention or control group (balanced randomization [1:1 ratio] based on computer-generated permutated blocks). Participants in the intervention group are required not to receive any other psychological or psychopharmacological intervention at study entry and during the training. Participants in the control group are required not to receive any psychological or psychopharmacological intervention at study entry. However, they may or may not engage in any intervention over the study course (usual care). After completion of the study, they will have the opportunity to receive the same self-efficacy training as the intervention group.

Sample size calculations are based on the "weakest line" in the analyses: Any incident or recurrent mental disorder from entry to follow-up assessment in the intervention vs. control group. Calculations are based on data from the baseline and first follow-up assessment of the Early Developmental Stages of Psychopathology Study, a population-based study of adolescents and young adults from Germany. Based on meta-analytic evidence on indicated mental health prevention, the investigators expect the intervention group to improve from standardized self-efficacy scores below -1 to scores between -1 and -0.5. In the EDSP, 21% of those with baseline scores between -1 and -0.5 (~ intervention group) and 41% of those with baseline scores below -1 (~ control group) developed any incident anxiety, affective, or substance use disorder until follow-up (considering only individuals without psychopathology at baseline). With a statistical power of 0.9 and a dropout rate of 20% (from baseline to post and from post to follow-up, respectively), an incidence rate of 21% vs. 41% in the intervention vs. control group yields 189 individuals required per group at baseline (total N=378).

Because a 12-month follow-up period is a relatively short time frame to evidence group differences in onset rates of full-threshold mental disorders, also incident/recurrent sub-threshold disorders will be considered. Sub-threshold disorders are defined as disorders falling short of one diagnostic criterion (e.g., the time criterion). In these analyses, incidences of sub-threshold disorders not being present at the entry assessment will be additionally counted.

Data Exclusion/Missing Data To ensure response accuracy and validity, several control items will be embedded in the assessments. Observations will be excluded if accuracy scores are too low.

Full information maximum likelihood estimation and, if necessary, other imputation methods (e.g., multiple imputation) will be used to deal with missing data.

Analysis Data analyses will be performed using RStudio, Python, Stata, and Mplus. Data from the main assessment will be analyzed using linear (dimensional outcomes) and logistic (binary outcomes) regressions. To test whether outcome changes from baseline to post/follow-up vary by group, the difference in the respective outcome score (post/follow-up minus baseline) will be regressed on a group dummy (0=control, 1=intervention). To test whether the rates of incident/recurrent mental disorders from study entry to follow-up vary by group, the diagnostic outcome will be regressed on the group dummy. To test for clinically significant effects, changes in clinical features (e.g., symptom burden and impairment) due to the intervention will be additionally assessed using linear/logistic regressions. EMA data will be analyzed using multilevel analyses with measurement occasions (level 1) nested within persons (level 2). To test whether outcome changes from baseline to post/follow-up vary by group, the respective outcome will be simultaneously regressed on a time dummy (0=baseline, 1=post/follow-up), a group dummy (0=control, 1=intervention), and an interaction term (time*group). Furthermore, multilevel models will be used to capture time-lagged associations between contextual factors and outcome changes in daily life. For example, the effect of daily hassles on momentary fluctuations in state self-efficacy and psychopathological symptoms in the intervention vs. control group will be examined. Dimensional outcomes with non-normally distributed residuals will be log-transformed (log(x+1)). To allow for comparisons across different measures and groups, all dimensional outcomes will be standardized (M=0, SD=1) based on the pooled standard deviation in the intervention and control groups at baseline (to account for potential baseline group differences). Analyses will be adjusted for gender and age. The alpha level will be set at .05. The "BY" method will be used to correct for multiple testing of dependent hypotheses. Spillover effects will be tested using multilevel models with time-lagged effects. If the power requirements are met random intercept cross-lagged panel models will be used. As a manipulation check, the investigators will test whether participants of the intervention group first increase in the domain of self-efficacy they work on (health, social relationships, or education/work) but not in the other domains. For example, individuals working on their health-related self-efficacy are expected to first increase in their health-related self-efficacy but not in the other 2 domains.

ELIGIBILITY:
Inclusion Criteria:

1. age 18-30 years and
2. low scores (≤24) on the German version of the General Self-Efficacy Scale (i.e., more than one standard deviation (5.4) below the mean score of 29.4 in the German norm sample; The cutoff will be raised to scores below the mean of 29.4 (≤30) if not enough participants with low self-efficacy scores of ≤24 and without 12-month mental disorders are found and this leads to serious problems regarding the recruitment phase and the timeline of the project.
3. ability to participate in the course (German language proficiency, availability during the intervention period)

Exclusion Criteria:

1. 12-month anxiety, affective, or substance use disorder (excluding nicotine dependence)
2. current psychological/psychopharmacological intervention or treatment seeking for psychological problems
3. acute suicidality; Individuals who report acute suicidality will be withdrawn from the study and referred to treatment.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 378 (Estimated)
Dates: Start 2024-11-18 (Actual); Primary Completion 2026-04-20 (Estimated); Study Completion 2026-04-20 (Estimated)

PRIMARY OUTCOMES:
Change in general self-efficacy measured by the German version of the General Self-Efficacy Scale (GSE) | From baseline to post (approximately 8-10 weeks).
  Change in general self-efficacy from baseline to post in the intervention group compared to the control group. The baseline measurement is taken immediately before the course starts, and the post measurement is taken within two weeks after the course ends. The interval between the two measurements is approximately 8-10 weeks, depending on participant availability. The German version of the General Self-Efficacy Scale (GSE) will be used. Scores range from 10 to 40, with higher scores indicating greater self-efficacy.
Rates of incident DSM-5 mental disorders assessed by the SCID-CV. | From baseline to follow-up (approximately 14 months).
  Rates of incident DSM-5 mental disorders from baseline to follow-up in the intervention group compared to the control group. Assessments occur at baseline and follow-up (approximately 14 months apart). Diagnoses will be made using the Structured Clinical Interview for DSM-5 (SCID-CV), focusing on sections A, D, E, and F, while sub-treshold symptoms are also assessed.

SECONDARY OUTCOMES:
Change in dimensional psychopathological symptoms measured by the DSM-5 Cross-Cutting-Symptom-Measure. | From baseline to post (approximately 8-10 weeks).
  Changes in anxiety, anger, somatic symptoms, depression, and anger from baseline to post-assessment in the intervention group compared to the control group. Baseline is conducted after study inclusion and before the course starts, and post-assessment is conducted within two weeks after the course ends (approximately 8-10 weeks). Scores for each symptom range from 0 to 4, with higher scores indicating more severe symptoms.
Change in dimensional psychopathological symptoms measured by the DSM-5 Cross-Cutting-Symptom-Measure. | From baseline to follow-up (approximately 14 months).
  Changes in anxiety, anger, somatic symptoms, depression, and anger from baseline to follow-up in the intervention group compared to the control group. Baseline assessments occur after study inclusion, and follow-up assessments occur 12 months after the post-assessment (approximately 14 months apart).
Change in self-esteem measured by the German version of the Rosenberg Self-Esteem Scale. | From baseline to post (approximately 8-10 weeks) and to follow-up (approximately 14 months).
  Changes in self-esteem from baseline to post-assessment to follow-up in the intervention group compared to the control group. The Rosenberg Self-Esteem Scale scores range from 10 to 40, with higher scores indicating better self-esteem.
Change in perceived control measured by the German version of the Perceived Control Scale (IE-4). | From baseline to post (approximately 8-10 weeks) and to follow-up (approximately 14 months).
  Changes in perceived control from baseline to post-assessment in the intervention group compared to the control group. The Perceived Control Scale scores range from 4 to 20, with higher scores indicating greater perceived control.
Change in perceived social support measured by the German version of the Multidimensional Scale of Perceived Social Support (MSPSS). | From baseline to post (approximately 8-10 weeks) and to follow-up (approximately 14 months).
  Changes in perceived social support from baseline to post-assessment in the intervention group compared to the control group. The MSPSS scores range from 12 to 84, with higher scores indicating greater perceived social support.
Change in coping measured by the German version of the COPE Inventory (28 items). | From baseline to post (approximately 8-10 weeks) and to follow-up (approximately 14 months).
  Changes in coping skills from baseline to post-assessment in the intervention group compared to the control group. The COPE Inventory scores range from 28 to 112, with higher scores indicating more effective coping strategies.
Change in interpersonal competence measured by the German version of the Interpersonal Competence Questionnaire (ICQ-15). | From baseline to post (approximately 8-10 weeks) and to follow-up (approximately 14 months).
  Changes in interpersonal competence from baseline to post-assessment in the intervention group compared to the control group. The ICQ-15 scores range from 15 to 60, with higher scores indicating better interpersonal competence.
Change in work engagement measured by the German version of the Utrecht Work Engagement Scale (UWES-9). | From baseline to post (approximately 8-10 weeks) and to follow-up (approximately 14 months).
  Changes in work engagement from baseline to post-assessment in the intervention group compared to the control group. The UWES scores range from 9 to 54, with higher scores indicating higher work engagement.
Change in individual work performance measured by the German version of the Individual Work Performance Questionnaire (IWPQ-18). | From baseline to post (approximately 8-10 weeks) and to follow-up (approximately 14 months).
  Changes in work performance from baseline to post-assessment in the intervention group compared to the control group. The IWPQ scores range from 18 to 90, with higher scores indicating better individual work performance.

CONTACTS AND LOCATIONS:
Locations (1):
- Health and Medical University Potsdam, Potsdam, Brandenburg, Germany

IPD SHARING:
Plan to Share IPD: Yes
Data for individual publications will be shared on OSF.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: After the end of the study
Access Criteria: Everyone; no restrictions
URL: https://osf.io/zbj73/

REFERENCES:
- [Background] Abramson LY, Seligman ME, Teasdale JD. Learned helplessness in humans: critique and reformulation. J Abnorm Psychol. 1978 Feb;87(1):49-74. No abstract available. PMID 649856
- [Background] Asselmann E, Wittchen HU, Lieb R, Hofler M, Beesdo-Baum K. Does low coping efficacy mediate the association between negative life events and incident psychopathology? A prospective-longitudinal community study among adolescents and young adults. Epidemiol Psychiatr Sci. 2016 Apr;25(2):171-80. doi: 10.1017/S204579601500013X. Epub 2015 Feb 25. PMID 25712151
- [Background] Bandura, A. (1986). Social Foundations of Thought and Action. Prentice Hall.
- [Background] Beierlein, C., Kovaleva, A., Kemper, C. J., & Rammstedt, B. (2012). ASKU-Allgemeine Selbstwirksamkeit Kurzskala.
- [Background] Beesdo-Baum K, Knappe S, Asselmann E, Zimmermann P, Bruckl T, Hofler M, Behrendt S, Lieb R, Wittchen HU. The 'Early Developmental Stages of Psychopathology (EDSP) study': a 20-year review of methods and findings. Soc Psychiatry Psychiatr Epidemiol. 2015 Jun;50(6):851-66. doi: 10.1007/s00127-015-1062-x. Epub 2015 May 16. PMID 25982479
- [Background] Benjamini, Y., & Hochberg, Y. (1995). Controlling the false discovery rate: A practical and powerful approach to multiple testing. Journal of the Royal Statistical Society B, 57, 289-300.
- [Background] Bentler PM. Comparative fit indexes in structural models. Psychol Bull. 1990 Mar;107(2):238-46. doi: 10.1037/0033-2909.107.2.238. PMID 2320703
- [Background] Bresó, E., Schaufeli, W. B., & Salanova, M. (2011). Can a self-efficacy-based intervention decrease burnout, increase engagement, and enhance performance? A quasi-experimental study. Higher Education, 61, 339-355.
- [Background] Cieslak R, Benight CC, Rogala A, Smoktunowicz E, Kowalska M, Zukowska K, Yeager C, Luszczynska A. Effects of Internet-Based Self-Efficacy Intervention on Secondary Traumatic Stress and Secondary Posttraumatic Growth among Health and Human Services Professionals Exposed to Indirect Trauma. Front Psychol. 2016 Jul 4;7:1009. doi: 10.3389/fpsyg.2016.01009. eCollection 2016. PMID 27458407
- [Background] Conley CS, Shapiro JB, Kirsch AC, Durlak JA. A meta-analysis of indicated mental health prevention programs for at-risk higher education students. J Couns Psychol. 2017 Mar;64(2):121-140. doi: 10.1037/cou0000190. PMID 28277730
- [Background] Cuijpers P. Examining the effects of prevention programs on the incidence of new cases of mental disorders: the lack of statistical power. Am J Psychiatry. 2003 Aug;160(8):1385-91. doi: 10.1176/appi.ajp.160.8.1385. PMID 12900296
- [Background] Dalgleish T, Black M, Johnston D, Bevan A. Transdiagnostic approaches to mental health problems: Current status and future directions. J Consult Clin Psychol. 2020 Mar;88(3):179-195. doi: 10.1037/ccp0000482. PMID 32068421
- [Background] Hinz, A., Schumacher, J., Albani, C., Schmid, G., & Brähler, E. (2006). Bevölkerungsrepräsentative Normierung der Skala zur allgemeinen Selbstwirksamkeitserwartung. Diagnostica, 52, 26-32.
- [Background] Khantzian EJ. The self-medication hypothesis of substance use disorders: a reconsideration and recent applications. Harv Rev Psychiatry. 1997 Jan-Feb;4(5):231-44. doi: 10.3109/10673229709030550. PMID 9385000
- [Background] Luszczynska A, Tryburcy M, Schwarzer R. Improving fruit and vegetable consumption: a self-efficacy intervention compared with a combined self-efficacy and planning intervention. Health Educ Res. 2007 Oct;22(5):630-8. doi: 10.1093/her/cyl133. Epub 2006 Oct 23. PMID 17060349
- [Background] Maciejewski PK, Prigerson HG, Mazure CM. Self-efficacy as a mediator between stressful life events and depressive symptoms. Differences based on history of prior depression. Br J Psychiatry. 2000 Apr;176:373-8. doi: 10.1192/bjp.176.4.373. PMID 10827887
- [Background] Muthén, L. K., & Muthén, B. O. (2017). Mplus: Statistical Analysis with Latent Variables: User's Guide (Version 8).
- [Background] Schonfeld P, Brailovskaia J, Bieda A, Zhang XC, Margraf J. The effects of daily stress on positive and negative mental health: Mediation through self-efficacy. Int J Clin Health Psychol. 2016 Jan-Apr;16(1):1-10. doi: 10.1016/j.ijchp.2015.08.005. Epub 2015 Oct 30. PMID 30487845
- [Background] Seligman ME. Learned helplessness. Annu Rev Med. 1972;23:407-12. doi: 10.1146/annurev.me.23.020172.002203. No abstract available. PMID 4566487
- [Background] StataCorp. (2021). Stata Statistical Software: Release 17.
- [Background] Volz M, Voelkle MC, Werheid K. General self-efficacy as a driving factor of post-stroke depression: A longitudinal study. Neuropsychol Rehabil. 2019 Oct;29(9):1426-1438. doi: 10.1080/09602011.2017.1418392. Epub 2018 Jan 4. PMID 29299953
- [Background] Wittchen HU, Knappe S, Andersson G, Araya R, Banos Rivera RM, Barkham M, Bech P, Beckers T, Berger T, Berking M, Berrocal C, Botella C, Carlbring P, Chouinard G, Colom F, Csillag C, Cujipers P, David D, Emmelkamp PM, Essau CA, Fava GA, Goschke T, Hermans D, Hofmann SG, Lutz W, Muris P, Ollendick TH, Raes F, Rief W, Riper H, Tossani E, van der Oord S, Vervliet B, Haro JM, Schumann G. The need for a behavioural science focus in research on mental health and mental disorders. Int J Methods Psychiatr Res. 2014 Jan;23 Suppl 1(Suppl 1):28-40. doi: 10.1002/mpr.1409. PMID 24375534
- See also: Study website — https://selftie-studie.de/